CLINICAL TRIAL: NCT05663307
Title: The Effect of Ginkgolide on Clinical Improvement of Patients With Acute Ischemic: A Randomized, Double Blind, Placebo Parallel Controlled Clinical Study
Brief Title: The Effect of Ginkgolide on Clinical Improvement of Patients With Acute Ischemic Stroke
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: No.2020-134
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Ischemic Stroke, Acute
MeSH Terms: conditions — Ischemic Stroke | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ginkgo diterpene lactone meglumine injection (Active Comparator): Intravenous injections of Ginkgo diterpene lactone meglumine injection at a dose of 25 mg (5ml) diluted with 250 ml physiological saline for 14 days ;Aspirin at a dose of 100 mg per day for 90 days.
  Interventions: Drug: Ginkgo diterpene lactone meglumine injection; Drug: Aspirin
- Ginkgo diterpene lactone meglumine injection simulation (Placebo Comparator): Intravenous injections of Ginkgo diterpene lactone meglumine injection simulation at a dose of 25 mg (5ml) diluted with 250 ml physiological saline for 14 days ;Aspirin at a dose of 100 mg per day for 90 days.
  Interventions: Drug: Ginkgo diterpene lactone meglumine injection simulation; Drug: Aspirin

INTERVENTIONS:
Drug: Ginkgo diterpene lactone meglumine injection — Intravenous injections of Ginkgo diterpene lactone meglumine injection at a dose of 25 mg (5ml) diluted with 250 ml physiological saline for 14 days plus aspirin at a dose of 100 mg per day for 90 days.
  Other Names: YinxingErtieneizhiPu'an Zhusheye
  Arms: Ginkgo diterpene lactone meglumine injection
Drug: Ginkgo diterpene lactone meglumine injection simulation — Intravenous injections of Ginkgo diterpene lactone meglumine injection simulation at a dose of 25 mg (5ml) diluted with 250 ml physiological saline for 14 days plus aspirin at a dose of 100 mg per day for 90 days.
  Other Names: YinxingErtieneizhiPu'an Zhusheye simulation
  Arms: Ginkgo diterpene lactone meglumine injection simulation
Drug: Aspirin — plus aspirin at a dose of 100 mg per day for 90 days.
  Other Names: Acetylsalicylic acid

SUMMARY:
The aim of this study is to evaluate the safety and effectivity of Ginkgo diterpene lactone meglumine injection tn the treatment of acute ischemic stroke

DETAILED DESCRIPTION:
This trial is a randomized, double-blind, placebo-controlled trial, A total of approximately 80 patients (age > 40 years) with acute ischemic stroke (5<NIHSS < 25), who can be treated within 4.5 to 48 hours of symptom onset will be enrolled. Patients fulfilling all of the inclusion criteria and none of the exclusion criteria will be randomized 1:1 into two groups after offering informed content: 1) one group will receive a Ginkgo Diterpene Lactone Meglumine Injection 25mg/5ml,once/day from Day 1 to Day 14（the injection must be added slowly into 0.9% sodium chloride injection diluted to 250 ml , intravenous drip for about 2 hours）, combined with Acetylsalicylic acid (Aspirin) at a dose of 100 mg/d for 90 days;2) the other group will receive the same volume saline injection as placebo for 14 days plus aspirin at a dose of 100 mg per day for 90 days.The primary objective is to assess the anti-platelet effects of Ginkgo Diterpene Lactone Meglumine Injection combined with Aspirin versus Aspirin alone in patients with acute ischemic stroke. The study consists of 3 visits including the day of randomization, Day 14±2days and Day 90±7days.After randomized to 90 + 7 days mRS 0-1 points is the Primary Outcome Measure,evaluate the safety and effectivity of Ginkgo diterpene lactone meglumine injection tn the treatment of acute ischemic stroke.A Data and Safety Monitoring Board (DSMB) will regularly monitor safety during the study. The trial has been approved by Ethics Committee of Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of Traditional Chinese Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 40 years, and gender not limited;
* Within 48 hours of stroke onset of ischemic stroke;
* The first onset, or always not obvious legacy of stroke sequela;
* A score of 5-24 points on the National Institute of Health Stroke Scale (NIHSS)；
* Understand and voluntarily signed informed consent.

Exclusion Criteria:

* Cardiogenic cerebral embolism;
* AIS caused by other definite causes (e.g., arterial dissection, vasculitis, vascular malformation, etc.) or undetermined etiology;
* Treated with thrombolysis or intravascular therapy, or with arteriovenous bridging after onset;
* Under dual antiplatelet therapy or anticoagulant therapy;
* A score of more than 2 on the modified Rankin Scale (mRS) (scores range from 0 [no symptoms] to 6 [death]) before the occurrence of AIS;
* Allergy or contraindication to GDLI or aspirin;
* Patients with active bleeding or bleeding tendency, malignancies, severe liver (the serum level of AST and/or ALT > 2 times the upper limit of normal), or renal failure (the serum level of creatinine > 1.5 times the upper limit of normal or GFR < 40 ml/min/1.73m2);
* Anticipated requirement for long-term nonstudy antiplatelet drugs or for nonsteroidal anti-inflammatory drugs affecting platelet function;
* Severe noncardiovascular coexisting condition, with a life expectancy of less than 3 months;
* Planned surgery or interventional treatment requiring cessation of the study drug;
* Pregnancy, lactation, or planning to get pregnant.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Modified Rankin Scale (mRS) | 90 days
  Proportion of patients with Modified Rankin Scale (mRS) less than or equal to 1 . The mRS scores range from 0 to 6, ranging from perfect health without symptoms to death

SECONDARY OUTCOMES:
New vascular events defined as any event of the following: Any stroke (ischemic or hemorrhage) | 90 days
  All the new vascular events will be assessed by at least two neurologists based on neuroimaging and clinical feature. When there was disagreement, a third senior neurologist was consulted to reach a consensus decision.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Han, Ph.D., Study Director — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Yueyang Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai University of Traditional Chinese Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No